CLINICAL TRIAL: NCT02425098
Title: A Phase II, Double-Blind, Randomized, Controlled Trial to Assess the Safety and Immunogenicity of a Tetravalent Dengue Vaccine With Two Different Serotype 2 Potencies in an Adult Population in Singapore
Brief Title: Safety and Immunogenicity With Two Different Serotype 2 Potencies of Takeda's Tetravalent Dengue Vaccine Candidate (TDV) in Adults in Singapore
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEN-205; U1111-1166-8884 (Registry Identifier: WHO)
Record Dates: First submitted 2015-04-09; First posted 2015-04-23 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Dengue Fever
Keywords: Vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose Tetravalent Dengue Vaccine (HD-TDV) (Experimental): High-dose Tetravalent Dengue Vaccine [HD-TDV], 0.5 mL, subcutaneous injection on Day 1. TDV comprised one molecularly-characterized and cloned TDV-2 live attenuated dengue virus strain and three recombinant live attenuated dengue virus strains: TDV-1, TDV-3 and TDV-4. TDV contained 2*10^4 plaque forming units (PFU), 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU of TDV-1, TDV-2, TDV-3 and TDV-4 respectively.
  Interventions: Biological: Takeda's High-Dose Tetravalent Dengue Vaccine Candidate (HD-TDV)
- Tetravalent Dengue Vaccine (TDV) (Experimental): Tetravalent Dengue Vaccine [TDV], 0.5 mL, subcutaneous injection on Day 1. TDV comprised one molecularly-characterized and cloned TDV-2 live attenuated dengue virus strain and three recombinant live attenuated dengue virus strains: TDV-1, TDV-3 and TDV-4. TDV contained 2*10^4 plaque forming units (PFU), 5*10^3 PFU, 1*10^5 PFU, and 3*10^5 PFU of TDV-1, TDV-2, TDV-3 and TDV-4 respectively.
  Interventions: Biological: Takeda's Tetravalent Dengue Vaccine Candidate (TDV)

INTERVENTIONS:
Biological: Takeda's Tetravalent Dengue Vaccine Candidate (TDV) — TDV subcutaneous injection
  Arms: Tetravalent Dengue Vaccine (TDV)
Biological: Takeda's High-Dose Tetravalent Dengue Vaccine Candidate (HD-TDV) — High-dose TDV subcutaneous injection
  Arms: High-dose Tetravalent Dengue Vaccine (HD-TDV)

SUMMARY:
The purpose of this study is to assess the post-vaccination neutralizing antibody response against each dengue serotype by vaccine group.

DETAILED DESCRIPTION:
The vaccine being tested in this study was Takeda's Tetravalent Dengue Vaccine Candidate (TDV). TDV is being tested to protect people against dengue fever. This study looked at safety and the titers of antibodies to dengue fever induced in people who were administered a high-dose of TDV (HD-TDV) compared to TDV.

The study enrolled 351 patients. Before being assigned to a treatment group participants were screened for previous exposure to the dengue virus using a Dengue immunoglobulin G (IgG) enzyme-linked immunosorbent assay (ELISA). Participants were randomly assigned in 1:1 ratio (by chance) to one of the two treatment groups-which remained undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* HD-TDV 0.5 mL subcutaneous injection
* TDV 0.5 mL subcutaneous injection

All participants received a single injection on Day 1. Participants were asked to record any symptoms that may or may not be related to the vaccine or the injection site in a diary card for 28 days after vaccination.

This multi-center trial was conducted in Singapore. The overall time of participation in this study was 12 months. Participants made multiple visits to the clinic, including a final visit 1 year after receiving their dose of TDV.

ELIGIBILITY:
Inclusion Criteria:

1. Participant signs and dates a written informed consent form where applicable, and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.
2. Is aged 21 to 45 years of age, inclusive.
3. Is in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the Investigator.
4. Can comply with trial procedures and are available for the duration of follow-up.
5. Has self-declared as never having been vaccinated against Yellow Fever or Japanese Encephalitis Virus.

Exclusion Criteria:

1. Has febrile illness (temperature ≥38°C or ≥100.4°F) or moderate or severe acute illness or infection at the time of enrollment.
2. Has history or any illness that, in the opinion of the Investigator, might interfere with the results of the trial or pose an additional risk to the participant due to participation in the trial, including but not limited to:

   1. Known hypersensitivity or allergy to any of the vaccine components.
   2. Female participants who are pregnant or breastfeeding.
   3. Individuals with any serious chronic or progressive disease according to judgment of the Investigator (e.g. neoplasm, insulin-dependent diabetes, cardiac, renal or hepatic disease, neurologic or seizure disorder or Guillain-Barré syndrome).
   4. Known or suspected impairment/alteration of immune function, including:

      * i. Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (Month 0) (use of inhaled, intranasal, or topical corticosteroids is allowed).
      * ii. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥ 2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (Month 0).
      * iii. Administration of immunoglobulins and/or any blood products within the 3 months prior to Day 1 (Month 0) or planned administration during the trial.
      * iv. Receipt of immunostimulants within 60 days prior to Day 1(Month 0).
      * v. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (Month 0).
      * vi. Human immunodeficiency virus (HIV) infection and HIV-related diseases.
      * vii. Hepatitis C virus (HCV) infection.
      * viii. Genetic immunodeficiency.
3. Has received any other vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to Day 1 (Month 0) or planning to receive any vaccine within 28 days after Day 1 (Month 0).
4. Has participated in any clinical trial with another investigational product 30 days prior to Day 1 (Month 0) or intent to participate in another clinical trial at any time during the conduct of this trial.
5. Has previously participated in any clinical trial of a dengue candidate vaccine, or previous receipt of a dengue vaccine.
6. Is first-degree relative of individuals involved in trial conduct.
7. For females of childbearing potential who are sexually active, and who have not used any of the acceptable contraceptive methods for at least 2 months prior to Day 1 (Month 0).

   1. Of childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: bilateral tubal ligation (at least 1 year previously), bilateral oophorectomy (at least 1 year previously) or hysterectomy.
   2. Acceptable birth control methods are defined as one or more of the following:

      * i. Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring).
      * ii. Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse.
      * iii. Intrauterine device (IUD).
      * iv. Monogamous relationship with vasectomized partner (partner must have been vasectomized for at least six months prior to Day 1 [Month 0]).
8. Females of childbearing potential who are sexually active, and who refuse to use an acceptable contraceptive method from signing the informed consent up to 6 weeks post-vaccination.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 351 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (3):
- Singapore (3):
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800
- [Derived] White LJ, Young EF, Stoops MJ, Henein SR, Adams EC, Baric RS, de Silva AM. Defining levels of dengue virus serotype-specific neutralizing antibodies induced by a live attenuated tetravalent dengue vaccine (TAK-003). PLoS Negl Trop Dis. 2021 Mar 12;15(3):e0009258. doi: 10.1371/journal.pntd.0009258. eCollection 2021 Mar. PMID 33711074
- [Derived] Michlmayr D, Andrade P, Nascimento EJM, Parker A, Narvekar P, Dean HJ, Harris E. Characterization of the Type-Specific and Cross-Reactive B-Cell Responses Elicited by a Live-Attenuated Tetravalent Dengue Vaccine. J Infect Dis. 2021 Feb 3;223(2):247-257. doi: 10.1093/infdis/jiaa346. PMID 32572472
- [Derived] Tricou V, Low JG, Oh HM, Leo YS, Kalimuddin S, Wijaya L, Pang J, Ling LM, Lee TH, Brose M, Hutagalung Y, Rauscher M, Borkowski A, Wallace D. Safety and immunogenicity of a single dose of a tetravalent dengue vaccine with two different serotype-2 potencies in adults in Singapore: A phase 2, double-blind, randomised, controlled trial. Vaccine. 2020 Feb 5;38(6):1513-1519. doi: 10.1016/j.vaccine.2019.11.061. Epub 2019 Dec 13. PMID 31843269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites into Singapore from 03 June 2015 to 18 September 2017.
Pre-assignment Details: Healthy volunteers were enrolled and randomized in 1:1 ratio to receive single injection of either high-dose tetravalent dengue vaccine (HD-TDV) or tetravalent dengue vaccine (TDV).
Period: Overall Study
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Started | 176 | 175
Completed | 163 | 159
Not Completed | 13 | 16
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Pregnancy | 2 | 0
Not completed — Reason not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all randomized participants who received the study vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV) | Total
Number analyzed (Participants) | 176 | 175 | 351
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (6.52) | 30.9 (6.74) | 31.0 (6.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 91 | 194
  Male | 73 | 84 | 157
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic or Latino | 176 | 175 | 351
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 173 | 172 | 345
  White | 1 | 2 | 3
  Multiracial | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 176 | 175 | 351
Height [Mean (Standard Deviation); unit: cm] | 164.26 (9.714) | 164.33 (9.505) | 164.29 (9.597)
Weight [Mean (Standard Deviation); unit: kg] | 66.44 (16.184) | 64.96 (16.295) | 65.70 (16.234)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI= (baseline weight in kg)/[(height in cm)/100]^2
  kg/m^2 | 24.51 (5.049) | 23.86 (4.681) | 24.18 (4.873)
Baseline Seropositivity Status [Count of Participants; unit: Participants] — Population: Data is reported only for participants with baseline seropositivity status.
  Participants
    Seropositive for at least one Dengue Serotype: number analyzed (Participants) | 175 | 175 | 350
    Seropositive for at least one Dengue Serotype | 92 | 95 | 187
    Seronegative for all Dengue Serotypes: number analyzed (Participants) | 175 | 175 | 350
    Seronegative for all Dengue Serotypes | 83 | 80 | 163
Baseline Seropositivity Rate for Each Serotype [Number; unit: percentage of participants] — Baseline seropositivity rate for each serotype is defined as percentage of participants seropositive for the given dengue serotype. Population: Participants with only seropositivity are reported.
  percentage of participants
    DENV-1: number analyzed (Participants) | 175 | 175 | 350
    DENV-1 | 48.6 | 48.6 | 48.6
    DENV-2: number analyzed (Participants) | 175 | 175 | 350
    DENV-2 | 47.4 | 50.3 | 48.9
    DENV-3: number analyzed (Participants) | 175 | 175 | 350
    DENV-3 | 44.0 | 46.3 | 45.1
    DENV-4: number analyzed (Participants) | 175 | 175 | 350
    DENV-4 | 41.7 | 40.6 | 41.1

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Neutralizing Antibody Titer (GMT) for Each of the Four Dengue Serotypes at Day 15
Description: GMTs were assessed for the four dengue serotypes: DENV-1, DENV-2, DENV-3, and DENV-4, by microneutralization test [MNT].
Time Frame: Day 15
Population: Per-protocol set (PPS) included all randomized participants who received study vaccine and for whom valid pre-dosing and at least one valid post-dosing MNT result was available, and who had no major protocol violations. Here 'number analyzed' refers to participants with valid MNT results available at given time-point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
Titer
  DENV-1: number analyzed (Participants) | 170 | 170
  DENV-1 | 156.2 [98.0 to 249.1] | 110.2 [73.8 to 164.6]
  DENV-2: number analyzed (Participants) | 170 | 170
  DENV-2 | 183.0 [116.7 to 287.0] | 117.6 [75.8 to 182.4]
  DENV-3: number analyzed (Participants) | 170 | 170
  DENV-3 | 113.5 [74.7 to 172.6] | 69.0 [47.1 to 100.9]
  DENV-4: number analyzed (Participants) | 170 | 170
  DENV-4 | 41.2 [29.7 to 57.2] | 33.9 [25.3 to 45.4]

2. Primary Outcome: Geometric Mean Neutralizing Antibody Titer (GMT) for Each of the Four Dengue Serotypes at Day 30
Description: GMTs were assessed for the four dengue serotypes: DENV-1, DENV-2, DENV-3, and DENV-4, by MNT.
Time Frame: Day 30
Population: The PPS included all randomized participants who received the study vaccine and for whom valid pre-dosing and at least one valid post-dosing MNT result was available, and who had no major protocol violations. Here 'number analyzed' refers to participants with valid MNT results available at given time-point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
Titer
  DENV-1: number analyzed (Participants) | 173 | 172
  DENV-1 | 771.0 [525.1 to 1132.0] | 470.5 [324.4 to 682.4]
  DENV-2: number analyzed (Participants) | 173 | 172
  DENV-2 | 8640.3 [7157.0 to 10431.0] | 1992.7 [1334.5 to 2975.5]
  DENV-3: number analyzed (Participants) | 173 | 172
  DENV-3 | 390.6 [262.1 to 582.2] | 250.8 [168.9 to 372.5]
  DENV-4: number analyzed (Participants) | 173 | 172
  DENV-4 | 110.2 [78.3 to 155.2] | 143.3 [107.0 to 191.8]

3. Primary Outcome: Geometric Mean Neutralizing Antibody Titer (GMT) for Each of the Four Dengue Serotypes at Day 90
Description: GMTs were assessed for the four dengue serotypes: DENV-1, DENV-2, DENV-3, and DENV-4, by MNT.
Time Frame: Day 90
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
Titer
  DENV-1: number analyzed (Participants) | 169 | 162
  DENV-1 | 376.5 [246.8 to 574.3] | 394.0 [265.0 to 585.9]
  DENV-2: number analyzed (Participants) | 169 | 162
  DENV-2 | 4090.2 [3439.8 to 4863.6] | 1647.3 [1158.5 to 2342.4]
  DENV-3: number analyzed (Participants) | 169 | 162
  DENV-3 | 266.5 [177.6 to 399.9] | 218.0 [148.1 to 320.8]
  DENV-4: number analyzed (Participants) | 169 | 162
  DENV-4 | 85.6 [61.7 to 118.6] | 117.4 [87.2 to 158.1]

4. Primary Outcome: Geometric Mean Neutralizing Antibody Titer (GMT) for Each of the Four Dengue Serotypes at Day 180
Description: GMTs were assessed for the four dengue serotypes: DENV-1, DENV-2, DENV-3, and DENV-4, by MNT.
Time Frame: Day 180
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
Titer
  DENV-1: number analyzed (Participants) | 166 | 163
  DENV-1 | 379.4 [252.3 to 570.3] | 312.2 [212.2 to 459.2]
  DENV-2: number analyzed (Participants) | 166 | 163
  DENV-2 | 2585.5 [2088.8 to 3200.3] | 1235.0 [890.7 to 1712.5]
  DENV-3: number analyzed (Participants) | 166 | 163
  DENV-3 | 236.2 [162.2 to 344.0] | 161.0 [110.5 to 234.6]
  DENV-4: number analyzed (Participants) | 166 | 163
  DENV-4 | 91.0 [65.7 to 125.9] | 92.9 [68.9 to 125.4]

5. Primary Outcome: Geometric Mean Neutralizing Antibody Titer (GMT) for Each of the Four Dengue Serotypes at Day 365
Description: GMTs were assessed for the four dengue serotypes: DENV-1, DENV-2, DENV-3, and DENV-4, by MNT.
Time Frame: Day 365
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
Titer
  DENV-1: number analyzed (Participants) | 160 | 156
  DENV-1 | 247.3 [160.9 to 380.2] | 264.1 [181.1 to 385.1]
  DENV-2: number analyzed (Participants) | 160 | 156
  DENV-2 | 1726.0 [1392.6 to 2139.3] | 809.5 [576.6 to 1136.4]
  DENV-3: number analyzed (Participants) | 160 | 156
  DENV-3 | 163.2 [110.0 to 242.3] | 132.6 [89.9 to 195.5]
  DENV-4: number analyzed (Participants) | 160 | 156
  DENV-4 | 75.3 [53.8 to 105.4] | 77.0 [56.9 to 104.2]

6. Primary Outcome: Seropositivity Rate for Each of the Four Dengue Serotypes at Day 15
Description: Seropositivity rate was defined as the percentage of participants being seropositive, derived from titers of dengue-neutralizing antibodies. Seropositivity was defined as a reciprocal neutralizing titer ≥10 (for each serotype). Seropositivity rates were assessed for the four dengue serotypes: DENV-1, DENV-2, DENV-3, and DENV-4.
Time Frame: Day 15
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
percentage of participants
  DENV-1: number analyzed (Participants) | 170 | 170
  DENV-1 | 70.0 [62.5 to 76.8] | 72.4 [65.0 to 78.9]
  DENV-2: number analyzed (Participants) | 170 | 170
  DENV-2 | 74.1 [66.9 to 80.5] | 65.9 [58.2 to 73.0]
  DENV-3: number analyzed (Participants) | 170 | 170
  DENV-3 | 68.8 [61.3 to 75.7] | 62.4 [54.6 to 69.7]
  DENV-4: number analyzed (Participants) | 170 | 170
  DENV-4 | 57.6 [49.8 to 65.2] | 60.6 [52.8 to 68.0]

7. Primary Outcome: Seropositivity Rate for Each of the Four Dengue Serotypes at Day 30
Description: as for outcome 6
Time Frame: Day 30
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
percentage of participants
  DENV-1: number analyzed (Participants) | 173 | 172
  DENV-1 | 97.1 [93.4 to 99.1] | 91.3 [86.0 to 95.0]
  DENV-2: number analyzed (Participants) | 173 | 172
  DENV-2 | 98.8 [95.9 to 99.9] | 89.5 [84.0 to 93.7]
  DENV-3: number analyzed (Participants) | 173 | 172
  DENV-3 | 89.0 [83.4 to 93.3] | 83.7 [77.3 to 88.9]
  DENV-4: number analyzed (Participants) | 173 | 172
  DENV-4 | 78.0 [71.1 to 84.0] | 87.2 [81.3 to 91.8]

8. Primary Outcome: Seropositivity Rate for Each of the Four Dengue Serotypes at Day 90
Description: as for outcome 6
Time Frame: Day 90
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
percentage of participants
  DENV-1: number analyzed (Participants) | 169 | 162
  DENV-1 | 89.3 [83.7 to 93.6] | 89.5 [83.7 to 93.8]
  DENV-2: number analyzed (Participants) | 169 | 162
  DENV-2 | 99.4 [96.7 to 100.0] | 92.6 [87.4 to 96.1]
  DENV-3: number analyzed (Participants) | 169 | 162
  DENV-3 | 85.8 [79.6 to 90.7] | 86.4 [80.2 to 91.3]
  DENV-4: number analyzed (Participants) | 169 | 162
  DENV-4 | 76.9 [69.8 to 83.0] | 86.4 [80.2 to 91.3]

9. Primary Outcome: Seropositivity Rate for Each of the Four Dengue Serotypes at Day 180
Description: as for outcome 6
Time Frame: Day 180
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
percentage of participants
  DENV-1: number analyzed (Participants) | 166 | 163
  DENV-1 | 93.4 [88.5 to 96.6] | 89.6 [83.8 to 93.8]
  DENV-2: number analyzed (Participants) | 166 | 163
  DENV-2 | 98.2 [94.8 to 99.6] | 92.6 [87.5 to 96.1]
  DENV-3: number analyzed (Participants) | 166 | 163
  DENV-3 | 88.0 [82.0 to 92.5] | 82.2 [75.5 to 87.7]
  DENV-4: number analyzed (Participants) | 166 | 163
  DENV-4 | 78.9 [71.9 to 84.9] | 84.0 [77.5 to 89.3]

10. Primary Outcome: Seropositivity Rate for Each of the Four Dengue Serotypes at Day 365
Description: as for outcome 6
Time Frame: Day 365
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
percentage of participants
  DENV-1: number analyzed (Participants) | 160 | 156
  DENV-1 | 84.4 [77.8 to 89.6] | 89.7 [83.9 to 94.0]
  DENV-2: number analyzed (Participants) | 160 | 156
  DENV-2 | 98.8 [95.6 to 99.8] | 91.0 [85.4 to 95.0]
  DENV-3: number analyzed (Participants) | 160 | 156
  DENV-3 | 79.4 [72.3 to 85.4] | 77.6 [70.2 to 83.8]
  DENV-4: number analyzed (Participants) | 160 | 156
  DENV-4 | 72.5 [64.9 to 79.3] | 81.4 [74.4 to 87.2]

11. Secondary Outcome: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary Recorded) Following Vaccination by Severity
Description: Solicited local AEs (at injection site) were collected by participants using diary cards within 7 days after vaccination and included pain [Grade 0 (no pain), 1 (mild: no interference with daily activity), 2 (moderate: interference with daily activity with or without treatment) and 3 (severe: prevents daily activity with or without treatment)], erythema [Grade 0 (<25 mm), 1 (25 - ≤ 50 mm), 2 (>50 - ≤ 100 mm), 3 (> 100 mm)] and swelling [Grade 0 (<25 mm), 1 (25 - ≤ 50 mm), 2 (>50 - ≤ 100 mm), 3 (> 100 mm)].
Time Frame: Within 7 days after Vaccination
Population: The safety set included all randomized participants who received the study vaccine. Here 'number analyzed' is the number of participants with data available for analysis. Only categories for which there was at least 1 participant are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 176 | 175
Participants
  Pain, Any Severity: number analyzed (Participants) | 175 | 175
  Pain, Any Severity | 81 | 91
  Pain, Grade 1: number analyzed (Participants) | 175 | 175
  Pain, Grade 1 | 77 | 84
  Pain, Grade 2: number analyzed (Participants) | 175 | 175
  Pain, Grade 2 | 3 | 6
  Pain, Grade 3: number analyzed (Participants) | 175 | 175
  Pain, Grade 3 | 1 | 1
  Erythema, Any Severity: number analyzed (Participants) | 175 | 175
  Erythema, Any Severity | 19 | 27
  Erythema, Grade 1: number analyzed (Participants) | 175 | 175
  Erythema, Grade 1 | 18 | 21
  Erythema, Grade 2: number analyzed (Participants) | 175 | 175
  Erythema, Grade 2 | 1 | 6
  Swelling, Any Severity: number analyzed (Participants) | 175 | 175
  Swelling, Any Severity | 3 | 4
  Swelling, Grade 1: number analyzed (Participants) | 175 | 175
  Swelling, Grade 1 | 3 | 4

12. Secondary Outcome: Number of Participants With Solicited Systemic Adverse Events (AEs) (Diary Recorded) Following Vaccination by Severity
Description: Solicited systemic AEs were collected by participants using diary cards within 14 days after vaccination and included fever, headache, asthenia, malaise and myalgia. Severity grades were: Grade 0: none, Grade 1: mild (no interference with daily activity), Grade 2: moderate (interference with daily activity with or without treatment), Grade 3: severe (prevents normal daily activity with or without treatment). A systemic AE of fever (defined as ≥ 100.4°F) was derived from a daily temperature reading recorded within 14 days after vaccination.
Time Frame: Within 14 days after Vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 176 | 175
Participants
  Headache, Any Severity: number analyzed (Participants) | 175 | 175
  Headache, Any Severity | 50 | 61
  Headache, Grade 1: number analyzed (Participants) | 175 | 175
  Headache, Grade 1 | 33 | 40
  Headache, Grade 2: number analyzed (Participants) | 175 | 175
  Headache, Grade 2 | 14 | 18
  Headache, Grade 3: number analyzed (Participants) | 175 | 175
  Headache, Grade 3 | 3 | 3
  Myalgia, Any Severity: number analyzed (Participants) | 175 | 175
  Myalgia, Any Severity | 47 | 47
  Myalgia, Grade 1: number analyzed (Participants) | 175 | 175
  Myalgia, Grade 1 | 38 | 33
  Myalgia, Grade 2: number analyzed (Participants) | 175 | 175
  Myalgia, Grade 2 | 7 | 11
  Myalgia, Grade 3: number analyzed (Participants) | 175 | 175
  Myalgia, Grade 3 | 2 | 3
  Asthenia, Any Severity: number analyzed (Participants) | 175 | 175
  Asthenia, Any Severity | 43 | 56
  Asthenia, Grade 1: number analyzed (Participants) | 175 | 175
  Asthenia, Grade 1 | 27 | 38
  Asthenia, Grade 2: number analyzed (Participants) | 175 | 175
  Asthenia, Grade 2 | 15 | 15
  Asthenia, Grade 3: number analyzed (Participants) | 175 | 175
  Asthenia, Grade 3 | 1 | 3
  Malaise, Any Severity: number analyzed (Participants) | 175 | 175
  Malaise, Any Severity | 41 | 49
  Malaise, Grade 1: number analyzed (Participants) | 175 | 175
  Malaise, Grade 1 | 26 | 32
  Malaise, Grade 2: number analyzed (Participants) | 175 | 175
  Malaise, Grade 2 | 12 | 12
  Malaise, Grade 3: number analyzed (Participants) | 175 | 175
  Malaise, Grade 3 | 3 | 5
  Fever, Any Severity: number analyzed (Participants) | 175 | 175
  Fever, Any Severity | 9 | 9
  Fever, 38.0-<38.5 (C): number analyzed (Participants) | 175 | 175
  Fever, 38.0-<38.5 (C) | 5 | 3
  Fever, 38.5-<39.0 (C): number analyzed (Participants) | 175 | 175
  Fever, 38.5-<39.0 (C) | 2 | 4
  Fever, 39.0-<39.5 (C): number analyzed (Participants) | 175 | 175
  Fever, 39.0-<39.5 (C) | 1 | 2
  Fever, 39.5-<40.0 (C): number analyzed (Participants) | 175 | 175
  Fever, 39.5-<40.0 (C) | 1 | 0

13. Secondary Outcome: Number of Participants With at Least One Unsolicited Adverse Events (AEs) Following Vaccination
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a study vaccine; it does not necessarily have to have a causal relationship with study vaccine administration.
Time Frame: Within 28 days after Vaccination
Population: The safety set included all randomized participants who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 176 | 175
Participants | 70 | 78

14. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above-mentioned criteria.
Time Frame: From first vaccination through end of study (Day 365)
Population: The safety set included all randomized participants who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 176 | 175
Participants | 3 | 3

15. Secondary Outcome: Geometric Mean Neutralizing Antibody Titers (GMT) for Each of the Four Dengue Serotypes Assessed by Dengue Baseline Seropositivity (MNT) Status
Description: Baseline dengue seropositivity was based on the microneutralization test (MNT) result and was defined as a reciprocal neutralizing titer ≥10 for one or more dengue serotype at baseline. The four DENV serotypes are DENV-1, DENV-2, DENV-3, and DENV-4.
Time Frame: Days 15, 30, 90, 180 and 365
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
Titer
  Day 15, DENV-1 (Seropositive): number analyzed (Participants) | 91 | 93
  Day 15, DENV-1 (Seropositive) | 1256.2 [734.1 to 2149.4] | 675.2 [441.2 to 1033.4]
  Day 15, DENV-2 (Seropositive): number analyzed (Participants) | 91 | 93
  Day 15, DENV-2 (Seropositive) | 1603.0 [1019.3 to 2521.1] | 1057.4 [699.4 to 1598.9]
  Day 15, DENV-3 (Seropositive): number analyzed (Participants) | 91 | 93
  Day 15, DENV-3 (Seropositive) | 677.7 [417.1 to 1101.0] | 376.0 [245.1 to 576.8]
  Day 15, DENV-4 (Seropositive): number analyzed (Participants) | 91 | 93
  Day 15, DENV-4 (Seropositive) | 181.8 [124.2 to 266.1] | 110.6 [78.8 to 155.1]
  Day 15, DENV-1 (Seronegative): number analyzed (Participants) | 79 | 77
  Day 15, DENV-1 (Seronegative) | 14.2 [10.3 to 19.4] | 12.3 [9.3 to 16.4]
  Day 15, DENV-2 (Seronegative): number analyzed (Participants) | 79 | 77
  Day 15, DENV-2 (Seronegative) | 15.0 [11.1 to 20.4] | 8.3 [6.8 to 10.2]
  Day 15, DENV-3 (Seronegative): number analyzed (Participants) | 79 | 77
  Day 15, DENV-3 (Seronegative) | 14.5 [10.3 to 20.4] | 8.9 [7.0 to 11.3]
  Day 15, DENV-4 (Seronegative): number analyzed (Participants) | 79 | 77
  Day 15, DENV-4 (Seronegative) | 7.5 [6.1 to 9.1] | 8.1 [6.3 to 10.4]
  Day 30, DENV-1 (Seropositive): number analyzed (Participants) | 91 | 94
  Day 30, DENV-1 (Seropositive) | 4058.9 [2651.9 to 6212.2] | 1763.7 [1168.7 to 2661.6]
  Day 30, DENV-2 (Seropositive): number analyzed (Participants) | 91 | 94
  Day 30, DENV-2 (Seropositive) | 6970.3 [5324.8 to 9124.3] | 4193.3 [3109.2 to 5655.5]
  Day 30, DENV-3 (Seropositive): number analyzed (Participants) | 91 | 94
  Day 30, DENV-3 (Seropositive) | 1940.7 [1242.3 to 3031.6] | 1015.7 [651.9 to 1582.7]
  Day 30, DENV-4 (Seropositive): number analyzed (Participants) | 91 | 94
  Day 30, DENV-4 (Seropositive) | 492.8 [342.8 to 708.5] | 304.7 [221.0 to 420.2]
  Day 30, DENV-1 (Seronegative): number analyzed (Participants) | 82 | 78
  Day 30, DENV-1 (Seronegative) | 122.0 [84.9 to 175.4] | 95.7 [61.0 to 150.1]
  Day 30, DENV-2 (Seronegative): number analyzed (Participants) | 82 | 78
  Day 30, DENV-2 (Seronegative) | 10965.9 [8472.9 to 14192.5] | 812.9 [376.0 to 1757.3]
  Day 30, DENV-3 (Seronegative): number analyzed (Participants) | 82 | 78
  Day 30, DENV-3 (Seronegative) | 65.9 [42.9 to 101.4] | 46.5 [29.0 to 74.6]
  Day 30, DENV-4 (Seronegative): number analyzed (Participants) | 82 | 78
  Day 30, DENV-4 (Seronegative) | 20.9 [14.9 to 29.3] | 57.7 [37.1 to 89.7]
  Day 90, DENV-1 (Seropositive): number analyzed (Participants) | 89 | 87
  Day 90, DENV-1 (Seropositive) | 2486.8 [1594.1 to 3879.3] | 1714.5 [1145.9 to 2565.1]
  Day 90, DENV-2 (Seropositive): number analyzed (Participants) | 89 | 87
  Day 90, DENV-2 (Seropositive) | 5501.1 [4473.6 to 6764.7] | 3601.4 [2626.0 to 4939.1]
  Day 90, DENV-3 (Seropositive): number analyzed (Participants) | 89 | 87
  Day 90, DENV-3 (Seropositive) | 1582.8 [1061.9 to 2359.3] | 925.6 [603.3 to 1420.1]
  Day 90, DENV-4 (Seropositive): number analyzed (Participants) | 89 | 87
  Day 90, DENV-4 (Seropositive) | 375.6 [267.7 to 526.9] | 303.8 [224.2 to 411.8]
  Day 90, DENV-1 (Seronegative): number analyzed (Participants) | 80 | 75
  Day 90, DENV-1 (Seronegative) | 46.1 [31.4 to 67.7] | 71.6 [43.7 to 117.1]
  Day 90, DENV-2 (Seronegative): number analyzed (Participants) | 80 | 75
  Day 90, DENV-2 (Seronegative) | 2941.4 [2243.1 to 3857.2] | 664.9 [360.3 to 1227.1]
  Day 90, DENV-3 (Seronegative): number analyzed (Participants) | 80 | 75
  Day 90, DENV-3 (Seronegative) | 36.7 [24.0 to 56.1] | 40.7 [26.5 to 62.7]
  Day 90, DENV-4 (Seronegative): number analyzed (Participants) | 80 | 75
  Day 90, DENV-4 (Seronegative) | 16.5 [12.3 to 22.2] | 39.0 [25.6 to 59.3]
  Day 180, DENV-1 (Seropositive): number analyzed (Participants) | 89 | 88
  Day 180, DENV-1 (Seropositive) | 2327.2 [1550.4 to 3493.3] | 1356.2 [905.5 to 2031.2]
  Day 180, DENV-2 (Seropositive): number analyzed (Participants) | 89 | 88
  Day 180, DENV-2 (Seropositive) | 4412.0 [3586.6 to 5427.4] | 2952.0 [2358.2 to 3695.4]
  Day 180, DENV-3 (Seropositive): number analyzed (Participants) | 89 | 88
  Day 180, DENV-3 (Seropositive) | 1248.3 [879.7 to 1771.3] | 693.6 [459.6 to 1046.6]
  Day 180, DENV-4 (Seropositive): number analyzed (Participants) | 89 | 88
  Day 180, DENV-4 (Seropositive) | 399.5 [291.3 to 547.9] | 268.3 [190.2 to 378.6]
  Day 180, DENV-1 (Seronegative): number analyzed (Participants) | 77 | 75
  Day 180, DENV-1 (Seronegative) | 46.6 [32.0 to 67.9] | 55.7 [35.6 to 87.1]
  Day 180, DENV-2 (Seronegative): number analyzed (Participants) | 77 | 75
  Day 180, DENV-2 (Seronegative) | 1394.1 [983.2 to 1976.6] | 444.3 [247.2 to 798.5]
  Day 180, DENV-3 (Seronegative): number analyzed (Participants) | 77 | 75
  Day 180, DENV-3 (Seronegative) | 34.5 [23.4 to 50.7] | 29.0 [19.4 to 43.3]
  Day 180, DENV-4 (Seronegative): number analyzed (Participants) | 77 | 75
  Day 180, DENV-4 (Seronegative) | 16.4 [12.3 to 22.0] | 26.8 [19.0 to 37.7]
  Day 365, DENV-1 (Seropositive): number analyzed (Participants) | 84 | 85
  Day 365, DENV-1 (Seropositive) | 1633.3 [1055.8 to 2526.7] | 1081.5 [724.0 to 1615.6]
  Day 365, DENV-2 (Seropositive): number analyzed (Participants) | 84 | 85
  Day 365, DENV-2 (Seropositive) | 3316.0 [2623.8 to 4190.9] | 2177.3 [1613.5 to 2938.1]
  Day 365, DENV-3 (Seropositive): number analyzed (Participants) | 84 | 85
  Day 365, DENV-3 (Seropositive) | 830.6 [551.2 to 1251.5] | 600.2 [402.3 to 895.3]
  Day 365, DENV-4 (Seropositive): number analyzed (Participants) | 84 | 85
  Day 365, DENV-4 (Seropositive) | 346.3 [249.2 to 481.1] | 212.6 [152.2 to 296.9]
  Day 365, DENV-1 (Seronegative): number analyzed (Participants) | 76 | 71
  Day 365, DENV-1 (Seronegative) | 30.7 [20.4 to 46.2] | 48.8 [32.1 to 74.2]
  Day 365, DENV-2 (Seronegative): number analyzed (Participants) | 76 | 71
  Day 365, DENV-2 (Seronegative) | 838.7 [621.9 to 1131.1] | 247.6 [143.9 to 426.1]
  Day 365, DENV-3 (Seronegative): number analyzed (Participants) | 76 | 71
  Day 365, DENV-3 (Seronegative) | 27.0 [17.8 to 41.1] | 21.7 [14.3 to 33.1]
  Day 365, DENV-4 (Seronegative): number analyzed (Participants) | 76 | 71
  Day 365, DENV-4 (Seronegative) | 13.9 [10.3 to 19.0] | 22.9 [15.8 to 33.1]

16. Secondary Outcome: Seropositivity Rate for Each of the Four Dengue Serotypes Assessed by Dengue Baseline Seropositivity (MNT) Status
Description: Baseline dengue seropositivity was based on the MNT result and was defined as a reciprocal neutralizing titer ≥10 for one or more dengue serotype at baseline. Seropositive rate was defined as a reciprocal neutralizing titer ≥ 10. Seropositivity was assessed for the four Dengue serotypes are DENV-1, DENV-2, DENV-3, and DEN-4.
Time Frame: Days 15, 30, 90, 180, and 365
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 173 | 174
percentage of participants
  Day 15, DENV-1 (Seropositive): number analyzed (Participants) | 91 | 93
  Day 15, DENV-1 (Seropositive) | 93.4 [86.2 to 97.5] | 98.9 [94.2 to 100.0]
  Day 15, DENV-2 (Seropositive): number analyzed (Participants) | 91 | 93
  Day 15, DENV-2 (Seropositive) | 93.4 [86.2 to 97.5] | 95.7 [89.4 to 98.8]
  Day 15, DENV-3 (Seropositive): number analyzed (Participants) | 91 | 93
  Day 15, DENV-3 (Seropositive) | 91.2 [83.4 to 96.1] | 91.4 [83.8 to 96.2]
  Day 15, DENV-4 (Seropositive): number analyzed (Participants) | 91 | 93
  Day 15, DENV-4 (Seropositive) | 89.0 [80.7 to 94.6] | 91.4 [83.8 to 96.2]
  Day 15, DENV-1 (Seronegative): number analyzed (Participants) | 79 | 77
  Day 15, DENV-1 (Seronegative) | 43.0 [31.9 to 54.7] | 40.3 [29.2 to 52.1]
  Day 15, DENV-2 (Seronegative): number analyzed (Participants) | 79 | 77
  Day 15, DENV-2 (Seronegative) | 51.9 [40.4 to 63.3] | 29.9 [20.0 to 41.4]
  Day 15, DENV-3 (Seronegative): number analyzed (Participants) | 79 | 77
  Day 15, DENV-3 (Seronegative) | 43.0 [31.9 to 54.7] | 27.3 [17.7 to 38.6]
  Day 15, DENV-4 (Seronegative): number analyzed (Participants) | 79 | 77
  Day 15, DENV-4 (Seronegative) | 21.5 [13.1 to 32.2] | 23.4 [14.5 to 34.4]
  Day 30, DENV-1 (Seropositive): number analyzed (Participants) | 91 | 94
  Day 30, DENV-1 (Seropositive) | 100.0 [96.0 to 100.0] | 100.0 [96.2 to 100.0]
  Day 30, DENV-2 (Seropositive): number analyzed (Participants) | 91 | 94
  Day 30, DENV-2 (Seropositive) | 98.9 [94.0 to 100.0] | 98.9 [94.2 to 100.0]
  Day 30, DENV-3 (Seropositive): number analyzed (Participants) | 91 | 94
  Day 30, DENV-3 (Seropositive) | 96.7 [90.7 to 99.3] | 95.7 [89.5 to 98.8]
  Day 30, DENV-4 (Seropositive): number analyzed (Participants) | 91 | 94
  Day 30, DENV-4 (Seropositive) | 94.5 [87.6 to 98.2] | 96.8 [91.0 to 99.3]
  Day 30, DENV-1 (Seronegative): number analyzed (Participants) | 82 | 78
  Day 30, DENV-1 (Seronegative) | 93.9 [86.3 to 98.0] | 80.8 [70.3 to 88.8]
  Day 30, DENV-2 (Seronegative): number analyzed (Participants) | 82 | 78
  Day 30, DENV-2 (Seronegative) | 98.8 [93.4 to 100.0] | 78.2 [67.4 to 86.8]
  Day 30, DENV-3 (Seronegative): number analyzed (Participants) | 82 | 78
  Day 30, DENV-3 (Seronegative) | 80.5 [70.3 to 88.4] | 69.2 [57.8 to 79.2]
  Day 30, DENV-4 (Seronegative): number analyzed (Participants) | 82 | 78
  Day 30, DENV-4 (Seronegative) | 59.8 [48.3 to 70.4] | 75.6 [64.6 to 84.7]
  Day 90, DENV-1 (Seropositive): number analyzed (Participants) | 89 | 87
  Day 90, DENV-1 (Seropositive) | 98.9 [93.9 to 100.0] | 100.0 [95.8 to 100.0]
  Day 90, DENV-2 (Seropositive): number analyzed (Participants) | 89 | 87
  Day 90, DENV-2 (Seropositive) | 100.0 [95.9 to 100.0] | 98.9 [93.8 to 100.0]
  Day 90, DENV-3 (Seropositive): number analyzed (Participants) | 89 | 87
  Day 90, DENV-3 (Seropositive) | 100.0 [95.9 to 100.0] | 97.7 [91.9 to 99.7]
  Day 90, DENV-4 (Seropositive): number analyzed (Participants) | 89 | 87
  Day 90, DENV-4 (Seropositive) | 95.5 [88.9 to 98.8] | 98.9 [93.8 to 100.0]
  Day 90, DENV-1 (Seronegative): number analyzed (Participants) | 80 | 75
  Day 90, DENV-1 (Seronegative) | 78.8 [68.2 to 87.1] | 77.3 [66.2 to 86.2]
  Day 90, DENV-2 (Seronegative): number analyzed (Participants) | 80 | 75
  Day 90, DENV-2 (Seronegative) | 98.8 [93.2 to 100.0] | 85.3 [75.3 to 92.4]
  Day 90, DENV-3 (Seronegative): number analyzed (Participants) | 80 | 75
  Day 90, DENV-3 (Seronegative) | 70.0 [58.7 to 79.7] | 73.3 [61.9 to 82.9]
  Day 90, DENV-4 (Seronegative): number analyzed (Participants) | 80 | 75
  Day 90, DENV-4 (Seronegative) | 56.3 [44.7 to 67.3] | 72.0 [60.4 to 81.8]
  Day 180, DENV-1 (Seropositive): number analyzed (Participants) | 89 | 88
  Day 180, DENV-1 (Seropositive) | 100.0 [95.9 to 100.0] | 100.0 [95.9 to 100.0]
  Day 180, DENV-2 (Seropositive): number analyzed (Participants) | 89 | 88
  Day 180, DENV-2 (Seropositive) | 100.0 [95.9 to 100.0] | 100.0 [95.9 to 100.0]
  Day 180, DENV-3 (Seropositive): number analyzed (Participants) | 89 | 88
  Day 180, DENV-3 (Seropositive) | 100.0 [95.9 to 100.0] | 96.6 [90.4 to 99.3]
  Day 180, DENV-4 (Seropositive): number analyzed (Participants) | 89 | 88
  Day 180, DENV-4 (Seropositive) | 95.5 [88.9 to 98.8] | 96.6 [90.4 to 99.3]
  Day 180, DENV-1 (Seronegative): number analyzed (Participants) | 77 | 75
  Day 180, DENV-1 (Seronegative) | 85.7 [75.9 to 92.6] | 77.3 [66.2 to 86.2]
  Day 180, DENV-2 (Seronegative): number analyzed (Participants) | 77 | 75
  Day 180, DENV-2 (Seronegative) | 96.1 [89.0 to 99.2] | 84.0 [73.7 to 91.4]
  Day 180, DENV-3 (Seronegative): number analyzed (Participants) | 77 | 75
  Day 180, DENV-3 (Seronegative) | 74.0 [62.8 to 83.4] | 65.3 [53.5 to 76.0]
  Day 180, DENV-4 (Seronegative): number analyzed (Participants) | 77 | 75
  Day 180, DENV-4 (Seronegative) | 59.7 [47.9 to 70.8] | 69.3 [57.6 to 79.5]
  Day 365, DENV-1 (Seropositive): number analyzed (Participants) | 84 | 85
  Day 365, DENV-1 (Seropositive) | 97.6 [91.7 to 99.7] | 100.0 [95.8 to 100.0]
  Day 365, DENV-2 (Seropositive): number analyzed (Participants) | 84 | 85
  Day 365, DENV-2 (Seropositive) | 100.0 [95.7 to 100.0] | 98.8 [93.6 to 100.0]
  Day 365, DENV-3 (Seropositive): number analyzed (Participants) | 84 | 85
  Day 365, DENV-3 (Seropositive) | 95.2 [88.3 to 98.7] | 96.5 [90.0 to 99.3]
  Day 365, DENV-4 (Seropositive): number analyzed (Participants) | 84 | 85
  Day 365, DENV-4 (Seropositive) | 95.2 [88.3 to 98.7] | 95.3 [88.4 to 98.7]
  Day 365, DENV-1 (Seronegative): number analyzed (Participants) | 76 | 71
  Day 365, DENV-1 (Seronegative) | 69.7 [58.1 to 79.8] | 77.5 [66.0 to 86.5]
  Day 365, DENV-2 (Seronegative): number analyzed (Participants) | 76 | 71
  Day 365, DENV-2 (Seronegative) | 97.4 [90.8 to 99.7] | 81.7 [70.7 to 89.9]
  Day 365, DENV-3 (Seronegative): number analyzed (Participants) | 76 | 71
  Day 365, DENV-3 (Seronegative) | 61.8 [50.0 to 72.8] | 54.9 [42.7 to 66.8]
  Day 365, DENV-4 (Seronegative): number analyzed (Participants) | 76 | 71
  Day 365, DENV-4 (Seronegative) | 47.4 [35.8 to 59.2] | 64.8 [52.5 to 75.8]

17. Secondary Outcome: Percentage of Participants Positive for Vaccine Viremia for Each of the Four Vaccine Strains After Vaccination
Description: Vaccine Viremia was assessed for each of the four vaccine strains: TDV-1, TDV-2, TDV-3 and TDV-4. Vaccine viral ribonucleic acid (RNA) was detected by reverse transcription-polymerase chain reaction (RT-PCR) assay.
Time Frame: Days 5, 7, 9, 11, 15, 17, 21 and 30
Population: Participants from the safety analysis set, all randomized participants who received at least 1 dose of study vaccine, with data available at the given time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 176 | 175
percentage of participants
  Day 5, TDV-1: number analyzed (Participants) | 172 | 174
  Day 5, TDV-1 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 5, TDV-2: number analyzed (Participants) | 172 | 174
  Day 5, TDV-2 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 5, TDV-3: number analyzed (Participants) | 172 | 174
  Day 5, TDV-3 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 5, TDV-4: number analyzed (Participants) | 172 | 174
  Day 5, TDV-4 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 7, TDV-1: number analyzed (Participants) | 175 | 174
  Day 7, TDV-1 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 7, TDV-2: number analyzed (Participants) | 175 | 174
  Day 7, TDV-2 | 16.6 [11.4 to 22.9] | 3.4 [1.3 to 7.4]
  Day 7, TDV-3: number analyzed (Participants) | 175 | 174
  Day 7, TDV-3 | 0.6 [0.0 to 3.1] | 0 [0.0 to 2.1]
  Day 7, TDV-4: number analyzed (Participants) | 175 | 174
  Day 7, TDV-4 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 9, TDV-1: number analyzed (Participants) | 168 | 172
  Day 9, TDV-1 | 0 [0.0 to 2.2] | 0 [0.0 to 2.1]
  Day 9, TDV-2: number analyzed (Participants) | 168 | 172
  Day 9, TDV-2 | 44.6 [37.0 to 52.5] | 13.4 [8.7 to 19.4]
  Day 9, TDV-3: number analyzed (Participants) | 168 | 172
  Day 9, TDV-3 | 0.6 [0.0 to 3.3] | 1.2 [0.1 to 4.1]
  Day 9, TDV-4: number analyzed (Participants) | 168 | 172
  Day 9, TDV-4 | 0 [0.0 to 2.2] | 0 [0.0 to 2.1]
  Day 11, TDV-1: number analyzed (Participants) | 171 | 172
  Day 11, TDV-1 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 11, TDV-2: number analyzed (Participants) | 171 | 172
  Day 11, TDV-2 | 48.0 [40.3 to 55.7] | 19.8 [14.1 to 26.5]
  Day 11, TDV-3: number analyzed (Participants) | 171 | 172
  Day 11, TDV-3 | 0 [0.0 to 2.1] | 0.6 [0.0 to 3.2]
  Day 11, TDV-4: number analyzed (Participants) | 171 | 172
  Day 11, TDV-4 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 15, TDV-1: number analyzed (Participants) | 172 | 171
  Day 15, TDV-1 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 15, TDV-2: number analyzed (Participants) | 172 | 171
  Day 15, TDV-2 | 35.5 [28.3 to 43.1] | 14.6 [9.7 to 20.8]
  Day 15, TDV-3: number analyzed (Participants) | 172 | 171
  Day 15, TDV-3 | 0.6 [0.0 to 3.2] | 0 [0.0 to 2.1]
  Day 15, TDV-4: number analyzed (Participants) | 172 | 171
  Day 15, TDV-4 | 0 [0.0 to 2.1] | 0.6 [0.0 to 3.2]
  Day 17, TDV-1: number analyzed (Participants) | 173 | 171
  Day 17, TDV-1 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 17, TDV-2: number analyzed (Participants) | 173 | 171
  Day 17, TDV-2 | 15.0 [10.1 to 21.2] | 11.7 [7.3 to 17.5]
  Day 17, TDV-3: number analyzed (Participants) | 173 | 171
  Day 17, TDV-3 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 17, TDV-4: number analyzed (Participants) | 173 | 171
  Day 17, TDV-4 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 21, TDV-1: number analyzed (Participants) | 175 | 172
  Day 21, TDV-1 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 21, TDV-2: number analyzed (Participants) | 175 | 172
  Day 21, TDV-2 | 0.6 [0.0 to 3.1] | 1.7 [0.4 to 5.0]
  Day 21, TDV-3: number analyzed (Participants) | 175 | 172
  Day 21, TDV-3 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 21, TDV-4: number analyzed (Participants) | 175 | 172
  Day 21, TDV-4 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 30, TDV-1: number analyzed (Participants) | 174 | 173
  Day 30, TDV-1 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 30, TDV-2: number analyzed (Participants) | 174 | 173
  Day 30, TDV-2 | 0 [0.0 to 2.1] | 0.6 [0.0 to 3.2]
  Day 30, TDV-3: number analyzed (Participants) | 174 | 173
  Day 30, TDV-3 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Day 30, TDV-4: number analyzed (Participants) | 174 | 173
  Day 30, TDV-4 | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]

18. Secondary Outcome: Duration of Vaccine Viremia for Each of the Four Vaccine Strains After Vaccination
Description: The duration of vaccine viremia for each vaccine strain was defined as the date when vaccine viremia was last detected (positive result) to date when vaccine viremia was first detected (positive result) + 1 day. It was assessed for each of the four vaccine strains: TDV-1, TDV-2, TDV-3 and TDV-4. Vaccine viral ribonucleic acid (RNA) was detected by reverse transcription-polymerase chain reaction (RT-PCR) assay.
Time Frame: Days 5, 7, 9, 11, 15, 17, 21 and 30
Population: Participants from the safety analysis set, all randomized participants who received at least 1 dose of study vaccine. Here 'number analyzed' refers to participants with a positive vaccine viremia test result.
Measure: Median (Full Range); unit: days
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 176 | 175
days
  TDV-1: number analyzed (Participants) | 0 | 0
  TDV-2: number analyzed (Participants) | 109 | 51
  TDV-2 | 5.0 [1 to 8] | 4.0 [1 to 10]
  TDV-3: number analyzed (Participants) | 3 | 3
  TDV-3 | 1.0 [1 to 1] | 1.0 [1 to 1]
  TDV-4: number analyzed (Participants) | 0 | 1
  TDV-4 |  | 1.0 [1 to 1]

19. Secondary Outcome: Level of Vaccine Viremia for Each of the Four Vaccine Strains After Vaccination
Description: as for outcome 17
Time Frame: Days 5, 7, 9, 11, 15, 17, 21 and 30
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: log10 [genome equivalents per mL]
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 176 | 175
log10 [genome equivalents per mL]
  Day 7, TDV-2: number analyzed (Participants) | 29 | 6
  Day 7, TDV-2 | 3.73 (0.631) | 3.78 (0.446)
  Day 7, TDV-3: number analyzed (Participants) | 1 | 0
  Day 7, TDV-3 | 2.82 (NA) — Standard Deviation (SD) was not calculated for 1 participant. |
  Day 9, TDV-2: number analyzed (Participants) | 75 | 23
  Day 9, TDV-2 | 3.63 (0.494) | 3.63 (0.711)
  Day 9, TDV-3: number analyzed (Participants) | 1 | 2
  Day 9, TDV-3 | 2.71 (NA) — SD was not calculated for 1 participant. | 2.67 (0.019)
  Day 11, TDV-2: number analyzed (Participants) | 82 | 34
  Day 11, TDV-2 | 3.64 (0.458) | 3.66 (0.481)
  Day 11, TDV-3: number analyzed (Participants) | 0 | 1
  Day 11, TDV-3 |  | 2.89 (NA) — SD was not calculated for 1 participant.
  Day 15, TDV-2: number analyzed (Participants) | 61 | 25
  Day 15, TDV-2 | 3.60 (0.320) | 3.54 (0.348)
  Day 15, TDV-3: number analyzed (Participants) | 1 | 0
  Day 15, TDV-3 | 2.81 (NA) — SD was not calculated for 1 participant. |
  Day 15, TDV-4: number analyzed (Participants) | 0 | 1
  Day 15, TDV-4 |  | 3.76 (NA) — SD was not calculated for 1 participant.
  Day 17, TDV-2: number analyzed (Participants) | 26 | 20
  Day 17, TDV-2 | 3.53 (0.336) | 3.44 (0.332)
  Day 21, TDV-2: number analyzed (Participants) | 1 | 3
  Day 21, TDV-2 | 3.57 (NA) — SD was not calculated for 1 participant. | 3.41 (0.426)
  Day 30, TDV-2: number analyzed (Participants) | 0 | 1
  Day 30, TDV-2 |  | 3.22 (NA) — SD was not calculated for 1 participant.

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: Within 28 days after Vaccination; SAEs: From first vaccination through end of study (Day 365)
Description: At each visit the investigator documented any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study vaccine.
Arm/Group | High-dose Tetravalent Dengue Vaccine (HD-TDV) | Tetravalent Dengue Vaccine (TDV)
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/175
Serious Adverse Events (participants affected / at risk) | 3/176 | 3/175
Other Adverse Events (participants affected / at risk) | 45/176 | 49/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Tetravalent Dengue Vaccine (HD-TDV) (N=176) | Tetravalent Dengue Vaccine (TDV) (N=175)
Retinal tear (Eye disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Barotrauma (Injury, poisoning and procedural complications) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Tetravalent Dengue Vaccine (HD-TDV) (N=176) | Tetravalent Dengue Vaccine (TDV) (N=175)
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 4 | 4
Injection site pruritus (General disorders) | 6 | 6
Vessel puncture site bruise (General disorders) | 4 | 8
Influenza (Infections and infestations) | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 6
Headache (Nervous system disorders) | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT02425098/SAP_000.pdf
  • Study Protocol (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT02425098/Prot_001.pdf